CLINICAL TRIAL: NCT00361946
Title: The Role of Amylin and Incretins on Postprandial Metabolisms in Adolescents With Type 2 Diabetes Mellitus (T2DM).
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Luisa M. Rodriguez, Senior Faculty, Baylor College of Medicine
Other Study IDs: NIH 1K126K63691; H-17370 (Other: BCM IRB)
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Lean; Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- lean subjects: BMI <85th for age, normal glucose tolerance
- obese subjects: BMI> 95th for age normal glucose tolerance
- Type diabetes: BMI > 85th for age , history of Type 2 diabetes as per ADA criteria

SUMMARY:
To study postprandial metabolism in lean, obese and T2DM adolescents using a mixed meal challenge. Specifically we will be measuring the following parameters of postprandial metabolism: 1. Postprandial glucose and triglycerides excursions 2. Gastric emptying 3. Insulin, amylin, glucagon, GLP-1 and ghrelin secretion 4. Glucose Turnover rate

DETAILED DESCRIPTION:
Previously type 2 diabetes mellitus (T2DM) was considered a disease of the adult; however, the incidence of T2DM in children is on the rise. Consequently, complications may occur at an earlier age, underscoring the importance of improving glycemic control in the pediatric population. Postprandial hyperglycemia contributes significantly to poor glycemic control in T2DM. We now understand that in addition to insulin other hormones (glucagon, amylin and GLP-1) may play a role in the postprandial glucose metabolism. The role of gastric emptying has been increasingly recognized as an important factor in regulating glucose appearance into the circulation. Abnormalities in the pancreatic hormone amylin and the incretin GLP-1 have emerged as contributors to the alterations in gastric emptying and postprandial hyperglycemia in T2DM. Although much is know about the abnormalities related to postprandial hyperglycemia in adults with T2DM, little information is available in the pediatric population. This protocol will examine gastric emptying, glucagon, GLP-1 and amylin secretions in healthy lean, obese children with and without diabetes post-ingestion of a mixed meal. The subject will be age and Tanner stage matched. The goal of this project is to better understand the metabolic adaptations of postprandial glucose homeostasis in T2DM by comparing our study group to obese (normal glucose tolerance) and healthy (lean) controls. The long-term goal for the PI is to use the data gathered with this protocol to develop a K-23 proposal incorporating new therapeutic options through the use of amylin and GLP-1 analogs in children with T2DM to improve postprandial hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Group A- Lean Adolescents a. Inclusion criteria: This group will consist of 20 lean adolescents between the ages of 12-18 years, Tanner stage 3-5 for pubertal development, have a BMI less than 85th and above 20th for age and an HbA1C less than or equal to 6% (normal range is 4-6%). They should not be taking any medications. A DXA scan will be performed to estimate lean and fat body mass. The body fat mass should be less than or equal to 25 % to be included in this group (in the lean range). The subjects will be matched for age and Tanner stage to the subjects in Group B and C. Menstruating females must have a negative urine pregnancy test for inclusion.The subject must weigh more than 43 kg.
2. Group B- Obese Adolescents a. Inclusion criteria: This group will consist of obese adolescents, between the ages of 12-18 years and Tanner stage 3-5 for pubertal development. They must have: a BMI above or equal to 95th for age, but not greater than 40 kg/m2 . They must have a normal glucose tolerance, in other words subjects with undiagnosed impaired glucose tolerance or diabetes will not be considered for the study. To test them for diabetes or impaired glucose tolerance they will undergo a 2-hour Glucose tolerance test (2hr-GTT). The ADA criteria will be used for the diagnosis of diabetes and/or impaired glucose tolerance (fasting plasma glucose < 110 mg/dl and a 2 hour postprandial blood glucose < 140 mg/dl). They must have and normal liver function tests and not taking any medications. The subjects will undergo DXA scan for estimation of total lean and fat body mass. The fat mass should be more than or equal to 30% to be considered obese. The subjects in this group will be matched for age (plus minus 1year), Tanner stage (plus minus 1) and body fat mass (plus minus 5%) to the Type 2 diabetes adolescents?. Menstruating females must have a negative urine pregnancy test for inclusion. 3. Group C- T2DM Adolescents a. Inclusion criteria The study group will consist of adolescents with T2DM, between the ages of 12-18 years, Tanner stage 3-5 for pubertal development, BMI above or equal to 85th for age (but less than 40 kg/m2) and HbA1c less than 8.5%. They must have T2DM diagnosed for at least 2years, treated with diet , oral hypoglycemic agents and or insulin. If on medications they need to be on a stable dose of insulin and / or oral hypoglycemic agent over the last 2 months. The subjects must be otherwise healthy except for hypothyroidism stable on treatment. Menstruating females must have a negative urine pregnancy test for inclusion. -

Exclusion Criteria:

1. Group A- Lean Adolescents a. Exclusion criteria: The subjects will be excluded if they have: a history of chronic disease (leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc), allergy to local anesthetics (ELAMAX Cream), evidence or history of chemical abuse, anemia and elevated liver enzymes (AST above 80 U/L and ALT above 110 U/L).
2. Group B- Obese Adolescents a. Exclusion criteria: The exclusion criteria are the same as for control group A.
3. Study Group C- T2DM Adolescents a. Exclusion Criteria: The exclusion criteria will be the same as in the control groups with one addition, subjects may not have been admitted to the hospital for diabetic ketoacidosis in the last 6 months.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents age 12-18
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa M Rodriguez, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided